CLINICAL TRIAL: NCT05329922
Title: Assistant for LIstening and Communication Enhancement
Acronym: ALICE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S66285
Record Dates: First submitted 2022-04-06; First posted 2022-04-15 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-08

CONDITIONS: Hearing Disability
Keywords: Auditory rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the training group or the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALICE (experienced hearing aid/cochlear implant users) (Experimental): Clients participating in this arm are asked to train their listening and communication skills using the ALICE app on their personal smart device for 8 weeks.
  Interventions: Behavioral: ALICE: Audiological rehabilitation
- Control (experienced hearing aid/cochlear implant users) (No Intervention): This arm will receive the standard of care given to the client. Persons with a moderate to profound hearing loss are provided with a hearing aid. Persons with a profound to severe HI are provided with a cochlear implant and concomitant rehabilitation. Most persons with a cochlear implant receive intensive rehabilitation during the first 6 months after their implantation. Afterwards, they mainly return for mapping of the device but not for listening training therapy.
- ALICE (new hearing aid users) (Experimental): Clients participating in this arm are asked to train their listening and communication skills using the ALICE app on their personal smart device during the hearing aid trial period (4-6 weeks on average).
  Interventions: Behavioral: ALICE: Audiological rehabilitation
- Control (new hearing aid users) (No Intervention): This arm will receive the standard of care given to the client during the hearing aid trial period.

INTERVENTIONS:
Behavioral: ALICE: Audiological rehabilitation — Persons who are randomised into this arm of the study will be asked to train their listening and communication skills using the ALICE app.
  Other Names: Use of the ALICE app
  Arms: ALICE (experienced hearing aid/cochlear implant users); ALICE (new hearing aid users)

SUMMARY:
As we get older, our hearing deteriorates and an age-related hearing loss can develop. Having a hearing loss can make it more difficult for people to understand conversations. Hearing aids can help in these situations, but difficulties often remain in more challenging situations, for example, when a conversation is being held in a group or when background noise is present. These difficulties are often not only related to the hearing loss but also to how these sounds are processed in the brain. Auditory rehabilitation is believed to help persons with a hearing impairment train their listening and communication skills. Auditory rehabilitation includes sensory management to enhance auditory function; knowledge and skills to improve the outcome; perceptual training and counselling. For this reason, the ALICE app was developed. The ALICE app contains monitoring tests, listening training exercises and counselling for persons with a hearing impairment.

In the current study, the ALICE app will be evaluated by persons with a hearing impairment. The experimental group will use the ALICE app in addition to the standard of care (hearing aid or cochlear implant) while the control group will receive the standard of care. Listening and communication skills will be evaluated pre and post training by a speech perception test in noise and questionnaires.

DETAILED DESCRIPTION:
This study is set-up as a pre-market clinical investigation of a non-CE marked medical device. The main goal of the study is to measure the efficacy of the ALICE app (Assistant for Listening and Communication Enhancement), a newly developed software application that will function as an added service in the aural rehabilitation of persons with HI, by providing remote monitoring, training and follow-up.

We will evaluate the efficacy and the clinical validity of the ALICE-app by means of a randomized controlled trial (RCT) with three arms. The first arm of the RCT will be carried out with 180 experienced hearing aid and/or cochlear implant users. The second arm of the RCT will be carried out with 120 first time hearing aid users. The third arm of the RCT includes an evaluation of the French version of the ALICE app, which will be carried out in 120 experienced hearing aid users from the French-speaking part of Belgium (the Walloon Region and Brussels).The participants will be divided in two groups: one group receiving the standard of care (control group), and another group receiving the standard of care supplemented with the ALICE-app.

All participants in the first and third arm will be assessed two times, at the beginning of the study and after 8 weeks of training (or without for the control group). The participants in the second arm will be assessed three times, at the beginning of the study, during the trial period with hearing aids and at the end of their trial period. The trial period with hearing aids takes on average 4-6 weeks. For the assessment we will use standardized clinical measures. These measures include a speech perception test in noise and validated questionnaires. The efficacy of ALICE will be determined in a within-subject design, i.e., baseline session outcomes will be compared to the final session outcomes of the randomized control trial, with a repeated measures ANOVA (α = 0.05).

ELIGIBILITY:
Inclusion Criteria (Experienced hearing aid/cochlear implant users):

* Clients with a hearing aid or cochlear implant.

  * Clients with a hearing aid must have completed the hearing aid trial period and must have decided to purchase the hearing aid.
  * Clients with a cochlear implant must have at least 6 months of experience with the implant.
* Clients who experience listening and communication difficulties.
* Clients may not have any experience with auditory training yet.
* Able to operate the training programme as an app on a mobile device/tablet (e.g. clients have a mobile device or table; clients have sufficient eyesight to see the exercises; clients must be able operate the programme).
* At least 18 years old.
* Arm 1: Dutch-speaking as all training material and counselling questions will be presented in Dutch.
* Arm 3: French-speaking as all training material and counselling questions will be presented in French.
* Clients need to have an Android or iPhone smart device and connection to internet

Inclusion Criteria (New hearing aid users):

* Clients who are starting their hearing aid trial as a first time hearing aid user (N= 120). Which is more than necessary according to the power analysis (3.5.7).
* Clients who experience listening and communication difficulties
* Able to operate the training programme as an app on a mobile device/tablet (e.g. clients have a mobile device or table; clients have sufficient eyesight to see the exercises; clients must be able operate the programme).
* At least 18 years old.
* Dutch-speaking as all training material and counselling questions will be presented in Dutch
* Clients need to have an Android or iPhone smartphone and connection to internet

Exclusion Criteria (Both groups):

* Visually impaired
* Motorically impaired
* Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2025-08-14 (Actual)

PRIMARY OUTCOMES:
Speech in noise intelligibility | During the first appointment before using the ALICE app
  Dutch: LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST, (van Wieringen & Wouters, 2008)) was specifically designed for speech perception in noise assessment in CI users. The test has a high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the ALICE app will be an improvement of 2dB on speech discrimination in noise.
  French: Listes disyllabiques de Lafon: disyllabic words presented in speech-weighted noise. Participants are required to repeat words in noise. The "Listes disyllabiques de Lafon" is a validated speech test during which French words are provided in quiet or in noise (Marie-Haps procedure).
Speech in noise intelligibility | After 8 weeks of training with the ALICE app during the final appointment
  Dutch: LIST (Leuven intelligibility sentences test) sentences presented in speech-weighted noise. Participants are required to repeat sentences in noise. The Leuven Intelligibility Sentences Test (LIST, (van Wieringen & Wouters, 2008)) was specifically designed for speech perception in noise assessment in CI users. The test has a high test-retest reliability and a steep slope making it very sensitive to small improvements in performance. An improvement of 2dB results in a clinically relevant improvement in speech discrimination in noise. Therefore, the primary endpoint to validate the ALICE app will be an improvement of 2dB on speech discrimination in noise.
  French: Listes disyllabiques de Lafon: disyllabic words presented in speech-weighted noise. Participants are required to repeat words in noise. The "Listes disyllabiques de Lafon" is a validated speech test during which French words are provided in quiet or in noise (Marie-Haps procedure).
Speech in noise intelligibility | During the first appointment before the hearing aid trial period
  BLU (Brugge-Leuven-Utrecht list) words presented in speech-weighted noise. Participants are required to repeat words in noise. The Brugge-Leuven-Utrecht list (BLU, ((Bosman, Woutes & Damman), 1994)) is a validated speech test during which Dutch words are provided in quiet or in noise. Each list contains 10 2-sylable words.
Speech in noise intelligibility | During an appointment 2 weeks into the hearing aid trial period
  BLU (Brugge-Leuven-Utrecht list) words presented in speech-weighted noise. Participants are required to repeat words in noise. The Brugge-Leuven-Utrecht list (BLU, ((Bosman, Woutes & Damman), 1994)) is a validated speech test during which Dutch words are provided in quiet or in noise. Each list contains 10 2-sylable words.
Speech in noise intelligibility | During the appointment at the end of the hearing aid trial period
  BLU (Brugge-Leuven-Utrecht list) words presented in speech-weighted noise. Participants are required to repeat words in noise. The Brugge-Leuven-Utrecht list (BLU, ((Bosman, Woutes & Damman), 1994)) is a validated speech test during which Dutch words are provided in quiet or in noise. Each list contains 10 2-sylable words.

SECONDARY OUTCOMES:
COSI (Client Oriented Scale of Improvement) | During the first appointment before using the ALICE app
  The COSI questionnaire is a validated clinical tool that can assist in measuring the impact of hearing aid fitting on a person's life and the benefit that is obtained after intervention (Dillon et al., 1997). Administering the COSI questionnaire is also part of the RIZIV/INAMI application to receive a refund for hearing aids. The COSI questionnaire allows the audiologist to measure improvements in listening situations important for their client. Before fitting the hearing aids, together with their client, they list their client's needs/goals. After hearing aids have been fitted and the client has had time to experience the hearing aids, they evaluate the progression/satisfaction in these situations together with their client.
COSI (Client Oriented Scale of Improvement) | During the first appointment before the hearing aid trial period
  The COSI questionnaire is a validated clinical tool that can assist in measuring the impact of hearing aid fitting on a person's life and the benefit that is obtained after intervention (Dillon et al., 1997). Administering the COSI questionnaire is also part of the RIZIV application to receive a refund for hearing aids. The COSI questionnaire allows the audiologist to measure improvements in listening situations important for their client. Before fitting the hearing aids, together with their client, they list their client's needs/goals. After hearing aids have been fitted and the client has had time to experience the hearing aids, they evaluate the progression/satisfaction in these situations together with their client.
COSI (Client Oriented Scale of Improvement) | After 8 weeks of training with the ALICE app during the final appointment
  The COSI questionnaire is a validated clinical tool that can assist in measuring the impact of hearing aid fitting on a person's life and the benefit that is obtained after intervention (Dillon et al., 1997). Administering the COSI questionnaire is also part of the RIZIV application to receive a refund for hearing aids. The COSI questionnaire allows the audiologist to measure improvements in listening situations important for their client. Before fitting the hearing aids, together with their client, they list their client's needs/goals. After hearing aids have been fitted and the client has had time to experience the hearing aids, they evaluate the progression/satisfaction in these situations together with their client.
COSI (Client Oriented Scale of Improvement) | During the appointment at the end of the hearing aid trial period
  The COSI questionnaire is a validated clinical tool that can assist in measuring the impact of hearing aid fitting on a person's life and the benefit that is obtained after intervention (Dillon et al., 1997). Administering the COSI questionnaire is also part of the RIZIV application to receive a refund for hearing aids. The COSI questionnaire allows the audiologist to measure improvements in listening situations important for their client. Before fitting the hearing aids, together with their client, they list their client's needs/goals. After hearing aids have been fitted and the client has had time to experience the hearing aids, they evaluate the progression/satisfaction in these situations together with their client.
CAS (Communication and Acceptance Scale) | During the first appointment before using the ALICE app
  The CAS is a validated scale that consist of 18 items (Öberg et al., 2021). The CAS scale is a reliable instrument that can be used to measure the effect of a rehabilitation programme. Each question is scored on a 5-point Likert scale (completely agree to completely disagree). It was developed to detect clinical changes in "communication strategies and the emotional consequences, knowledge and acceptance of hearing loss". This questionnaire has been translated from Swedish to Dutch and French (and back translated to ensure correct translation).
CAS (Communication and Acceptance Scale) | During the first appointment before the hearing aid trial period
  The CAS is a validated scale that consist of 18 items (Öberg et al., 2021). The CAS scale is a reliable instrument that can be used to measure the effect of a rehabilitation programme. Each question is scored on a 5-point Likert scale (completely agree to completely disagree). It was developed to detect clinical changes in "communication strategies and the emotional consequences, knowledge and acceptance of hearing loss". This questionnaire has been translated from Swedish to Dutch and French (and back translated to ensure correct translation).
CAS (Communication and Acceptance Scale) | During an appointment 2 weeks into the hearing aid trial period
  The CAS is a validated scale that consist of 18 items (Öberg et al., 2021). The CAS scale is a reliable instrument that can be used to measure the effect of a rehabilitation programme. Each question is scored on a 5-point Likert scale (completely agree to completely disagree). It was developed to detect clinical changes in "communication strategies and the emotional consequences, knowledge and acceptance of hearing loss". This questionnaire has been translated from Swedish to Dutch and French (and back translated to ensure correct translation).
CAS (Communication and Acceptance Scale) | After 8 weeks of training with the ALICE app during the final appointment
  The CAS is a validated scale that consist of 18 items (Öberg et al., 2021). The CAS scale is a reliable instrument that can be used to measure the effect of a rehabilitation programme. Each question is scored on a 5-point Likert scale (completely agree to completely disagree). It was developed to detect clinical changes in "communication strategies and the emotional consequences, knowledge and acceptance of hearing loss". This questionnaire has been translated from Swedish to Dutch and French (and back translated to ensure correct translation).
CAS (Communication and Acceptance Scale) | During the appointment at the end of the hearing aid trial period
  The CAS is a validated scale that consist of 18 items (Öberg et al., 2021). The CAS scale is a reliable instrument that can be used to measure the effect of a rehabilitation programme. Each question is scored on a 5-point Likert scale (completely agree to completely disagree). It was developed to detect clinical changes in "communication strategies and the emotional consequences, knowledge and acceptance of hearing loss". This questionnaire has been translated from Swedish to Dutch and French (and back translated to ensure correct translation).
EAS (Effort Assessment Scale) | During the first appointment before using the ALICE app
  EAS is a validated scale to measure listening effort (Alhanbali et al., 2017). The EAS consists of 6 items that are scored by the client on a 10-point scale, no effort to lots of effort. The EAS questions were translated to Dutch and French for this study.
EAS (Effort Assessment Scale) | After 8 weeks of training with the ALICE app during the final appointment
  EAS is a validated scale to measure listening effort (Alhanbali et al., 2017). The EAS consists of 6 items that are scored by the client on a 10-point scale, no effort to lots of effort. The EAS questions were translated to Dutch and French for this study.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | During the first appointment before using the ALICE app
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. (Noble et al., 2013). Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch and French.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | During the first appointment before the hearing aid trial period
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. (Noble et al., 2013). Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch and French.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | After 8 weeks of training with the ALICE app during the final appointment
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. (Noble et al., 2013). Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch and French.
SSQ12 (Speech, Spatial and Qualities of Hearing Scale) | During the appointment at the end of the hearing aid trial period
  The SSQ12 is a short version of the validated Speech, Spatial and Qualities of Hearing Scale. This short form was developed for use in clinical research and rehabilitation settings. (Noble et al., 2013). Participants score each questions on a ruler (visual analogue scale) from 0 to 10. Questions were translated to Dutch and French.
IOI-HA (International Outcome Inventory for Hearing Aids) | During the first appointment before using the ALICE app
  The IOI-HA (International Outcome Inventory for Hearing Aids) evaluates the daily use of the hearing aid, as well as the perceived benefit and satisfaction with the hearing aids or cochlear implants. The IOI-HA consist of 7 questions and has been validated in Dutch (Kramer et al., 2002).
IOI-HA (International Outcome Inventory for Hearing Aids) | During the first appointment before the hearing aid trial period
  The IOI-HA (International Outcome Inventory for Hearing Aids) evaluates the daily use of the hearing aid, as well as the perceived benefit and satisfaction with the hearing aids or cochlear implants. The IOI-HA consist of 7 questions and has been validated in Dutch (Kramer et al., 2002).
IOI-HA (International Outcome Inventory for Hearing Aids) | After 8 weeks of training with the ALICE app during the final appointment
  The IOI-HA (International Outcome Inventory for Hearing Aids) evaluates the daily use of the hearing aid, as well as the perceived benefit and satisfaction with the hearing aids or cochlear implants. The IOI-HA consist of 7 questions and has been validated in Dutch (Kramer et al., 2002).
IOI-HA (International Outcome Inventory for Hearing Aids) | During the appointment at the end of the hearing aid trial period
  The IOI-HA (International Outcome Inventory for Hearing Aids) evaluates the daily use of the hearing aid, as well as the perceived benefit and satisfaction with the hearing aids or cochlear implants. The IOI-HA consist of 7 questions and has been validated in Dutch (Kramer et al., 2002).
The ALICE-specific Questionnaire | During an appointment 2 weeks into the hearing aid trial period
  A specific ALICE-questionnaire was developed for the purpose of this study. The questions of this questionnaire were based on 3 different questionnaires. First, the SUS (system usability scale) to determine the usability of the ALICE app. Second, the SADL (Satisfaction with Amplification in Daily Living) which was designed to evaluate the satisfaction that people experience with their hearing aids. Third, the PREM (Patient Reported Experience Measures) as is used to evaluate audiological centres in the Netherlands. A total of 20 questions were selected to evaluate the participants' experience with the usability of the ALICE app, their satisfaction with their hearing aids and their satisfaction with their audiologist/hearing centre. The questionnaire is used in Dutch and French.
The ALICE-specific Questionnaire | During the appointment at the end of the hearing aid trial period
  A specific ALICE-questionnaire was developed for the purpose of this study. The questions of this questionnaire were based on 3 different questionnaires. First, the SUS (system usability scale) to determine the usability of the ALICE app. Second, the SADL (Satisfaction with Amplification in Daily Living) which was designed to evaluate the satisfaction that people experience with their hearing aids. Third, the PREM (Patient Reported Experience Measures) as is used to evaluate audiological centres in the Netherlands. A total of 20 questions were selected to evaluate the participants' experience with the usability of the ALICE app, their satisfaction with their hearing aids and their satisfaction with their audiologist/hearing centre.
  The questionnaire is used in Dutch and French.

CONTACTS AND LOCATIONS:
Overall Officials: Astrid van Wieringen, PhD, Principal Investigator — KU Leuven
Locations (1):
- KU Leuven, Experimental ORL, Dept Neurosciences, Leuven, VLAAMS BRABANT, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] van Wieringen A, Van Wilderode M, De Ridder L, Francart T, Wouters J. ALICE: Improved Speech in Noise Understanding with Self-guided Hearing Care. Trends Hear. 2025 Jan-Dec;29:23312165251393034. doi: 10.1177/23312165251393034. Epub 2025 Nov 10. PMID 41212721

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT05329922/Prot_SAP_000.pdf